CLINICAL TRIAL: NCT03637556
Title: A Multi-Center, Open-Label, Two-Period Cross-Over, Patient-Pilot Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Iron Chelating Activity of DST-0509 (Deferasirox) Tablets in Thalassemia Patients With Inadequate Response to Standard Chelation Therapy
Brief Title: Pilot Study to Assess the Safety, PK and Iron Chelating Activity of DST-0509 (Deferasirox) in Thalassemia Patients Refractory to Chelation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DisperSol Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DST-0509-201
Record Dates: First submitted 2018-07-30; First posted 2018-08-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Thalassemia Major
Keywords: thalassemia; iron; chelation; deferasirox; DST-0509; transfusion
MeSH Terms: conditions — beta-Thalassemia; Thalassemia | interventions — Deferasirox

STUDY DESIGN:
Intervention Model Description: open-label, two-period cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DST-0509 (Experimental): DST-0509 (deferasirox) will be supplied in 360 mg, 180 mg and 90 mg tablets. DST-0509 is taken once daily with food; the first dose will be taken at Visit 3 (Day 1) and the final dose will be taken at Visit 10 (Day 63).
  Interventions: Drug: DST-0509
- Jadenu (Active Comparator): Jadenu is commercially available as tablets and will be provided by the patient with their ongoing prescription. Dosing will be at equivalent (mg for mg) doses of DST-0509 or Jadenu. Jadenu is taken once daily with or without a light meal. However, Jadenu can be administered according to the patient's current prescription regimen. The first dose will be taken at Visit 3 (Day 1) and the final dose will be taken at Visit 10 (Day 63).
  Interventions: Drug: Jadenu
- Exjade (Active Comparator): Exjade is commercially available as tablets and Exjade as tablets for oral suspension and will be provided by the patient with their ongoing prescription. Dosing will be at equivalent (mg for mg) doses of DST-0509 or Jadenu. If converting from Exjade, the dose will be scaled for each treatment by 28 mg/40 mg (treatment/Exjade). Jadenu and Exjade are taken once daily, Jadenu is taken with or without a light meal, and Exjade is recommended to be taken without food. However, either Jadenu or Exjade can be administered according to the patient's current prescription regimen. The first dose will be taken at Visit 3 (Day 1) and the final dose will be taken at Visit 10 (Day 63).
  Interventions: Drug: Exjade

INTERVENTIONS:
Drug: DST-0509 — Novel iron chelator with improved absorption characteristics
  Other Names: deferasirox tablets
  Arms: DST-0509
Drug: Jadenu — Commercial iron chelator with standard absorption characteristics
  Other Names: deferasirox tablets
  Arms: Jadenu
Drug: Exjade — Commercial iron chelator with standard absorption characteristics
  Other Names: deferasirox oral suspension
  Arms: Exjade

SUMMARY:
This study is a multicenter, open-label, two-period crossover design that evaluates the safety, tolerability, pharmacokinetics and preliminary evidence of iron chelating activity of DST-0509 as compared to Jadenu and Exjade in transfusion-dependent thalassemia patients with transfusional iron overload, requiring iron chelation therapy and demonstrating an inadequate response to Jadenu or Exjade for greater than 3 months duration. Up to 36 patients will be evaluated (18 in each treatment arm), however, the balanced randomization may enroll fewer patients based on recruitment status.

DETAILED DESCRIPTION:
This is a multi-center, open-label, two-period cross-over, patient-pilot study comparing DST-0509 to patient's prior ICT (Exjade or Jadenu) administered orally once daily (QD) for 28-days in each period, with a 6-day washout before the first treatment period, between treatment periods, and at the end of the study before patients recommence their prescription regimens. Patients will be randomized to one of two treatment sequences: DST 0509→Exjade/Jadenu or Exjade/Jadenu→DST-0509 (with subjects who were taking Exjade prior to study start receiving Exjade and those taking Jadenu at study start receiving Jadenu). This study is designed to assess the safety, tolerability, evidence of iron chelating activity, and PK profile of DST-0509 compared to Jadenu or Exjade in inadequately responding patients.

Up to 36 patients will be randomized 1:1 into one of two treatment sequences (study arms), of which up to 100% may be on Jadenu or Exjade at study entry, or a mix of the two. The planned randomization will assign up to 18 patients in each of two sequences: Sequence A: DST-0509 crossed to Exjade or Jadenu; Sequence B: Jadenu or Exjade crossed to DST-0509. The comparator treatment will be the patient's current chelation treatment. At the end of the study, patients previously on Jadenu or Exjade will revert to receiving their pre-study medication and dose following a 6-day washout period. A sufficient number of patients will be enrolled so there will be no need to replace study drop-outs. Study duration is approximately 14 weeks for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent or assent as appropriate obtained prior to any study-related procedure being performed;
2. Patients at least 8 years of age or older at the time of consent or assent;
3. Patient with TDT syndrome and iron overload currently receiving iron chelation therapy with Jadenu or Exjade and demonstrating inadequate response assessed with serum ferritin and LIC;
4. At least 8 or more blood transfusions in the past year;
5. Survival expected of >12 months;
6. Patient previously on dual iron chelation therapy will be transfered to iron chelation monotherapy ,stable dosing with Jadenu or Exjade for ≥1month prior to screening and receiving doses in the maximal dose range per day (e.g., Jadenu: >21 mg/kg or Exjade: >30 mg/kg, with specific doses in these ranges prescribed at the physician's discretion);
7. Serum ferritin levels that are persistently >800 mcg/L determined by 2 separate assessments during screening over the previous 2-4 weeks prior to study treatment and not showing a decreasing trend over these weeks OR, an LIC of >5 mg Fe/g dw measured by MRI in the 52 weeks prior to study entry, OR clearly identified as a poor responder in medical records within 3 months prior to the study
8. Compliant with chelation therapy in the 3 months prior to enrollment in the opinion of the Investigator; has taken at least 75% of medication prescribed on a regular basis was taken (Investigator enquiry into patient prescription refill records, preferably 3 months if available, SICT scores); and

   1. Willing to comply with chelation therapy for the duration of the study;
   2. The determination of compliance is at the discretion of the investigator.
9. Agree not to use other anti-chelating agents concurrently;
10. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
11. Women of childbearing potential (WOCBP) must use an adequate method of birth control (double barrier, e.g. hormonal control and barrier contraception) at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug;
12. Male patients whose partners are WOCBP must use an adequate method of birth control (double barrier control) at least 28 days prior to the first administration of the study drug, during the study and for at least 30 days after the last dose of the study drug; and
13. Patient is willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria:

1. Females of childbearing potential not on an adequate method of birth control, or who are pregnant or lactating;
2. History of non-compliance with chelation therapy (determined by the investigator).
3. Known history of human immunodeficiency virus (HIV)
4. Active hepatitis B virus (HBV), hepatitis C virus (HCV), or other known active viral hepatitis;
5. Screening blood counts as follows:

   1. Absolute neutrophil count < 1,000/μL
   2. Platelets < 50,000/μL
   3. Hemoglobin < 7 g/dL (transfusion support is permitted);
6. Screening chemistry values as follows:

   1. Alanine aminotransferase (ALT) and aspartate transaminase (AST) > 3 × upper limit of the normal reference range (ULN)
   2. Total bilirubin > 5 × ULN
   3. Creatinine > 1.5 × ULN
   4. Urine protein/creatinine ratio (UPCR) > 0.5 mg/mg
   5. Albumin < 2.8 g/dL;
7. History of congestive heart failure New York Heart Association (NYHA) class III or IV or uncontrolled hypertension at screening;
8. History of other malignancy within the previous 3 years, except basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer;
9. In the opinion of the Investigator, evidence of major inflammatory disease that would affect ferritin levels within 14 days prior to the start of study medication;
10. Major surgery within 30 days prior to the start of study medication;
11. Serious persistent infection within 14 days prior to the start of study medication;
12. Serious concurrent medical condition including central nervous system (CNS) disorders;
13. Requires concomitant treatment with systemic corticosteroids, or any other immunosuppressive agents, or has used such treatment in the past 10 days before study entry (use of prednisone or equivalent <10 mg/day orally or use of inhaled corticosteroids or topical steroids is permitted);
14. Previous history of difficulty swallowing oral medications;
15. Any condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures or study medication; or
16. Concomitant treatment with medications described in Section "Prohibited Medications".

Patients who screen fail for out-of-protocol laboratory values may be re-screened at the Investigator's discretion provided that more than 30 days have passed since their previous screening. Up to three re-screenings will be permitted.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
diarrhea % | Up to Day 70
  safety tolerability
Ferritin (mcg/L) | Up to Day 63
  iron chelating activity

SECONDARY OUTCOMES:
Area Under the Curve (AUC), mg*h/L | Days 1, 7, 28, 36, 42 and 63
  Area Under the Plasma Curve
Maximum concentration (Cmax), mg/L | Days 1, 7, 28, 36, 42 and 63
  Peak exposure, Maximum plasma concentration
Time to maximum concentration (Tmax), h | Days 1, 7, 28, 36, 42 and 63
  Time to maximum plasma concentration.

CONTACTS AND LOCATIONS:
Locations (4):
- Weill Cornell Medicine, New York-Presbyterian Hospital, New York, New York, United States
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Thalassemia Center Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai